CLINICAL TRIAL: NCT07121920
Title: A Prospective Study Evaluating Ex-vivo Confocal Imaging of Fluorescent Tagged Monoclonal Antibodies and Proteomic Profiles of Biopsied Tissue to Predict Therapeutic Response Among Children and Adolescents With Inflammatory Bowel Disease
Brief Title: Ex-vivo Confocal Imaging and Proteomic Profiling to Determine Treatment Response in Children With IBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Children's Health Care System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-083
Record Dates: First submitted 2025-08-12; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: IBD (Inflammatory Bowel Disease); IBD; IBD - Inflammatory Bowel Disease
Keywords: Ex-vivo; Inflammatory bowel disease; IBD; CLE; Confocal laser endomicroscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Pediatric patients with clinical signs and symptoms suggestive of IBD or with established diagnosis of IBD (newly diagnosed or on therapeutic management) who are scheduled to undergo Esophagogastroduodenoscopy (EGD) and/or Ileocolonoscopy (IC) with CLE as part of their clinical management
  Interventions: Device: Confocal Laser Endomicroscopy

INTERVENTIONS:
Device: Confocal Laser Endomicroscopy — Patients will undergo Esophagogastroduodenoscopy (EGD) and/or Ileocolonoscopy (IC) EGD with CLE as per standard of care. Each participant will have 3-4 mucosal biopsies taken from the terminal ileum, rectosigmoid and cecum, ideally from the most affected areas of accessible segment.
  Ex vivo staining of biopsied tissue will be expanded to include FITC-labeled antibodies to cytokines IL12 and IL12/IL23 and to cytokine receptors IL12R and IL23R and possibly other cytokines, receptors and adhesion molecules. All biopsies tested for membrane bound antibodies will be done using CLE technology with artificial intelligence (AI). The cellular landscape will be characterized by surveying surface markers using bar-coded antibodies and performing gene expression profiling on every cell within inflamed tissue of patients with IBD.
  We will develop algorithm using AI to predict responders versus non-responders and to further subclassify IBD patients using phenotype data.

SUMMARY:
This study aims to test the overall hypothesis that the membrane tissue binding capacity of cytokines in the biopsied tissue of patients with Inflammatory Bowel Disease (IBD) is predictive of/strongly correlated to clinical response/outcomes observed.

The key questions under investigation are:

Aim 1: To assess the fluorescent signal intensity at baseline (control antibody with control biopsy and control antibody with IBD biopsy).

Aim 2: To characterize the cellular landscape by surveying surface markers using bar-coded antibodies and performing gene expression profiling on every cell within inflamed tissue of patients with IBD.

Aim 3: Develop algorithm using artificial intelligence to predict responders versus non-responders and to further subclassify IBD patients using phenotype data.

DETAILED DESCRIPTION:
It is estimated that approximately 5-10% of IBD patients develop the disease during childhood or adolescence. The disease onset peaks in adolescence, while 4% of children with IBD are less than 5 years of age and 18% below 10 years of age. IBD is characterized by a prolonged course of remission and relapse.

In patients with suspected IBD, endoscopy with biopsy is the gold standard method to diagnose and assess the degree and extent of inflammation. The impairment of intact intestinal epithelial barrier function is the hallmark of IBD, further involving a cascade of molecular and cellular alterations leading to delayed mucosal wound healing.

In the past decade, several studies examined the utility of probe-based confocal laser endomicroscopy (CLE) in several diseases, including IBD. The CLE is an emerging endoscopic technology developed to obtain high magnification and high-resolution images known as "optical" biopsies of the gastrointestinal mucosal histology in real-time at the cellular and sub-cellular levels.

The advantage of CLE during endoscopy is that normal tissue can be identified in real-time with high precision. A semi-quantitative test known as the Watson score was described by to describe structural and functional barrier defects in the terminal ileum in inflammatory bowel disease using CLE.

Although the use of biologics has revolutionized the management of IBD, it is estimated that approximately 10-40% of patients with IBD on biological agents like anti-TNF such as Infliximab (IFX) are primary non-responders, with an additional 13% per patient year experiencing a secondary loss of response. In children with moderate to severe Crohn's disease, it was estimated that only 67% would continue maintenance infliximab after three-years and approximately 50% of pediatric patients on IFX require dose intensification during maintenance therapy.

Limited studies have explored the binding of fluorescent labeled biologics ex-vivo using CLE in adults with little to no published literature in children. Studies in Europe have demonstrated that greater the binding of the biologic agent to the biopsied tissue pre-treatment, was associated with increased response to treatment, which was more pronounced in Ulcerative Colitis (AUROC 83%, PPV 89%, NPV 50%). A study abstract reported to have assessed the presence of fluorescein isothicyanate (FITC) labeled Vedolizumab (VDZ) prior to initiation of VDZ therapy in five patients with Crohn's Disease refractory to anti-TNF therapy. Among the 5, two of them showed α4β7 expressing mucosal cells and were found to have a good response to subsequent treatment with VDZ. However, further details of the study were not available. Similarly, a sustained improved response to anti-TNF treatment among patients with Crohn's Disease with high membrane-bound tumor necrosis factor (mTNF) intestinal immune cells using CLE evidenced by mucosal healing was observed on follow-up endoscopy compared to those who had low mTNF levels.

We sought to pursue the proposed study for the following reasons:

1. Unlike adults, IBD is more aggressive in children, for eg. impairs physical growth, impacting quality of life, in addition to the medication toxicities on top of the limited treatment options for IBD in pediatric patients.
2. The current approach in the management of IBD is treat to target, to achieve mucosal healing5 as subclinical inflammation could persist (as evidenced by endoscopy or histologically active disease) even though signs and symptoms have resolved. The above testing kit couples the use of CLE to determine treatment response, which aligns with the before-mentioned therapeutic goals in the management of IBD.
3. The cost of biologics are one of the major barriers to access of this promising treatment. At Cook Children's Health Care System, an average of 3-4 children/adolescents are diagnosed with Crohn's Disease or Ulcerative Colitis per week. Physicians can judiciously use biologics depending on treatment response assessed by the proposed testing kit, which will help alleviate the overall burden of cost incurred, to both the individual as well as to the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

- Patients must fall into one of the below categories: (i) with suspected and/or established diagnosis of IBD (ii) patients with IBD on treatment with biologics irrespective of treatment response (iii) patients who are diagnosed with IBD but treatment naïve to biologics. (iv) patients diagnosed with IBS and previous endoscopy results were negative for IBD who will serve as controls

Exclusion Criteria:

* Those with previous allergy to fluorescein
* Pregnant and breastfeeding patients

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of FITC tagged antibodies | Baseline
  Count of FITC tagged antibodies that maintain target specificity using fluorescence microplate reader. Used to establish baseline for fluorescent signal using FITC-tagged control antibody and control biopsy and IBD biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Huang, MD, Principal Investigator — Cook Children's Health Care System
Locations (2):
- United States (2):
  - University of Texas at Arlington, Arlington, Texas
  - Cook Children's Health Care System, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghione S, Sarter H, Fumery M, Armengol-Debeir L, Savoye G, Ley D, Spyckerelle C, Pariente B, Peyrin-Biroulet L, Turck D, Gower-Rousseau C, Andre JM, Antonietti M, Aouakli A, Armand A, Aroichane I, Assi F, Aubet JP, Auxenfants E, Ayafi-Ramelot F, Bankovski D, Barbry B, Bardoux N, Baron P, Baudet A, Bazin B, Bebahani A, Becqwort JP, Benet V, Benali H, Benguigui C, Soussan BE, Bental A, Berkelmans I, Bernet J, Bernou K, Bernou-Dron C, Bertot P, Bertiaux-Vandaele N, Bertrand V, Billoud E, Biron N, Bismuth B, Bleuet M, Blondel F, Blondin V, Bohon P, Boniface E, Bonniere P, Bonvarlet E, Bonvarlet P, Boruchowicz A, Bostvironnois R, Boualit M, Bouche B, Boudaillez C, Bourgeaux C, Bourgeois M, Bourguet A, Bourienne A, Branche J, Bray G, Brazier F, Breban P, Brihier H, Brung-Lefebvre V, Bulois P, Burgiere P, Butel J, Canva JY, Canva-Delcambre V, Capron JP, Cardot F, Carpentier P, Cartier E, Cassar JF, Cassagnou M, Castex JF, Catala P, Cattan S, Catteau S, Caujolle B, Cayron G, Chandelier C, Chantre M, Charles J, Charneau T, Chavance-Thelu M, Chirita D, Choteau A, Claerbout JF, Clergue PY, Coevoet H, Cohen G, Collet R, Colombel JF, Coopman S, Corvisart J, Cortot A, Couttenier F, Crinquette JF, Crombe V, Dadamessi I, Dapvril V, Davion T, Dautreme S, Debas J, Degrave N, Dehont F, Delatre C, Delcenserie R, Delette O, Delgrange T, Delhoustal L, Delmotte JS, Demmane S, Deregnaucourt G, Descombes P, Desechalliers JP, Desmet P, Desreumaux P, Desseaux G, Desurmont P, Devienne A, Devouge E, Devred M, Devroux A, Dewailly A, Dharancy S, Di Fiore A, Djeddi D, Djedir R, Dreher-Duwat ML, Dubois R, Dubuque C, Ducatillon P, Duclay J, Ducrocq B, Ducrot F, Ducrotte P, Dufilho A, Duhamel C, Dujardin D, Dumant-Forest C, Dupas JL, Dupont F, Duranton Y, Duriez A, El Achkar K, El Farisi M, Elie C, Elie-Legrand MC, Elkhaki A, Eoche M, Evrard D, Evrard JP, Fatome A, Filoche B, Finet L, Flahaut M, Flamme C, Foissey D, Fournier P, Foutrein-Comes MC, Foutrein P, Fremond D, Frere T, Fumery M, Gallet P, Gamblin C, Ganga-Zandzou PS, Gerard R, Geslin G, Gheyssens Y, Ghossini N, Ghrib S, Gilbert T, Gillet B, Godard D, Godard P, Godchaux JM, Godchaux R, Goegebeur G, Goria O, Gottrand F, Gower P, Grandmaison B, Groux M, Guedon C, Guillard JF, Guillem L, Guillemot F, Guimber D, Haddouche B, Hakim S, Hanon D, Hautefeuille V, Heckestweiller P, Hecquet G, Hedde JP, Hellal H, Henneresse PE, Heyman B, Heraud M, Herve S, Hochain P, Houssin-Bailly L, Houcke P, Huguenin B, Iobagiu S, Ivanovic A, Iwanicki-Caron I, Janicki E, Jarry M, Jeu J, Joly JP, Jonas C, Katherin F, Kerleveo A, Khachfe A, Kiriakos A, Kiriakos J, Klein O, Kohut M, Kornhauser R, Koutsomanis D, Laberenne JE, Laffineur G, Lagarde M, Lannoy P, Lapchin J, Lapprand M, Laude D, Leblanc R, Lecieux P, Leclerc N, Le Couteulx C, Ledent J, Lefebvre J, Lefiliatre P, Legrand C, Le Grix A, Lelong P, Leluyer B, Lenaerts C, Lepileur L, Leplat A, Lepoutre-Dujardin E, Leroi H, Leroy MY, Lesage JP, Lesage X, Lesage J, Lescanne-Darchis I, Lescut J, Lescut D, Leurent B, Levy P, Lhermie M, Lion A, Lisambert B, Loire F, Louf S, Louvet A, Luciani M, Lucidarme D, Lugand J, Macaigne O, Maetz D, Maillard D, Mancheron H, Manolache O, Marks-Brunel AB, Marti R, Martin F, Martin G, Marzloff E, Mathurin P, Mauillon J, Maunoury V, Maupas JL, Mesnard B, Metayer P, Methari L, Meurisse B, Meurisse F, Michaud L, Mirmaran X, Modaine P, Monthe A, Morel L, Mortier PE, Moulin E, Mouterde O, Mudry J, Nachury M, Khac NE, Notteghem B, Ollevier V, Ostyn A, Ouraghi A, Ouvry D, Paillot B, Panien-Claudot N, Paoletti C, Papazian A, Parent B, Pariente B, Paris JC, Patrier P, Paupart L, Pauwels B, Pauwels M, Petit R, Piat M, Piotte S, Plane C, Plouvier B, Pollet E, Pommelet P, Pop D, Pordes C, Pouchain G, Prades P, Prevost A, Prevost JC, Quesnel B, Queuniet AM, Quinton JF, Rabache A, Rabelle P, Raclot G, Ratajczyk S, Rault D, Razemon V, Reix N, Revillon M, Richez C, Robinson P, Rodriguez J, Roger J, Roux JM, Rudelli A, Saber A, Savoye G, Schlosseberg P, Segrestin M, Seguy D, Serin M, Seryer A, Sevenet F, Shekh N, Silvie J, Simon V, Spyckerelle C, Talbodec N, Techy A, Thelu JL, Thevenin A, Thiebault H, Thomas J, Thorel JM, Tielman G, Tode M, Toisin J, Tonnel J, Touchais JY, Touze Y, Tranvouez JL, Triplet C, Turck D, Uhlen S, Vaillant E, Valmage C, Vanco D, Vandamme H, Vanderbecq E, Eecken VE, Vandermolen P, Vandevenne P, Vandeville L, Vandewalle A, Vandewalle C, Vaneslander P, Vanhoove JP, Vanrenterghem A, Varlet P, Vasies I, Verbiese G, Vernier-Massouille G, Vermelle P, Verne C, Vezilier-Cocq P, Vigneron B, Vincendet M, Viot J, Voiment YM, Wacrenier A, Waeghemaecker L, Wallez JY, Wantiez M, Wartel F, Weber J, Willocquet JL, Wizla N, Wolschies E, Zalar A, Zaouri B, Zellweger A, Ziade C; Epimad Group. Dramatic Increase in Incidence of Ulcerative Colitis and Crohn's Disease (1988-2011): A Population-Based Study of French Adolescents. Am J Gastroenterol. 2018 Feb;113(2):265-272. doi: 10.1038/ajg.2017.228. Epub 2017 Aug 15. PMID 28809388
- [Background] Rath T, Bojarski C, Neurath MF, Atreya R. Molecular imaging of mucosal alpha4beta7 integrin expression with the fluorescent anti-adhesion antibody vedolizumab in Crohn's disease. Gastrointest Endosc. 2017 Aug;86(2):406-408. doi: 10.1016/j.gie.2017.01.012. Epub 2017 Jan 27. No abstract available. PMID 28137597
- [Background] Iacucci M, Jeffery L, Acharjee A, Grisan E, Buda A, Nardone OM, Smith SCL, Labarile N, Zardo D, Ungar B, Hunter S, Mao R, Cannatelli R, Shivaji UN, Parigi TL, Reynolds GM, Gkoutos GV, Ghosh S. Computer-Aided Imaging Analysis of Probe-Based Confocal Laser Endomicroscopy With Molecular Labeling and Gene Expression Identifies Markers of Response to Biological Therapy in IBD Patients: The Endo-Omics Study. Inflamm Bowel Dis. 2023 Sep 1;29(9):1409-1420. doi: 10.1093/ibd/izac233. PMID 36378498
- [Background] Hyams JS, Lerer T, Griffiths A, Pfefferkorn M, Kugathasan S, Evans J, Otley A, Carvalho R, Mack D, Bousvaros A, Rosh J, Mamula P, Kay M, Crandall W, Oliva-Hemker M, Keljo D, LeLeiko N, Markowitz J; Pediatric Inflammatory Bowel Disease Collaborative Research Group. Long-term outcome of maintenance infliximab therapy in children with Crohn's disease. Inflamm Bowel Dis. 2009 Jun;15(6):816-22. doi: 10.1002/ibd.20845. PMID 19107783
- [Background] Gisbert JP, Panes J. Loss of response and requirement of infliximab dose intensification in Crohn's disease: a review. Am J Gastroenterol. 2009 Mar;104(3):760-7. doi: 10.1038/ajg.2008.88. Epub 2009 Jan 27. PMID 19174781
- [Background] Rath T, Atreya R, Bodenschatz J, Uter W, Geppert CE, Vitali F, Fischer S, Waldner MJ, Colombel JF, Hartmann A, Neurath MF. Intestinal Barrier Healing Is Superior to Endoscopic and Histologic Remission for Predicting Major Adverse Outcomes in Inflammatory Bowel Disease: The Prospective ERIca Trial. Gastroenterology. 2023 Feb;164(2):241-255. doi: 10.1053/j.gastro.2022.10.014. Epub 2022 Oct 21. PMID 36279923
- [Background] Lim LG, Neumann J, Hansen T, Goetz M, Hoffman A, Neurath MF, Galle PR, Chan YH, Kiesslich R, Watson AJ. Confocal endomicroscopy identifies loss of local barrier function in the duodenum of patients with Crohn's disease and ulcerative colitis. Inflamm Bowel Dis. 2014 May;20(5):892-900. doi: 10.1097/MIB.0000000000000027. PMID 24691113
- [Background] Auzoux J, Boschetti G, Anon B, Aubourg A, Caulet M, Poisson L, Besson P, Lecomte T, Roger S, Picon L, Nancey S, Moussata D, Flourie B. Usefulness of confocal laser endomicroscopy for predicting postoperative recurrence in patients with Crohn's disease: a pilot study. Gastrointest Endosc. 2019 Jul;90(1):151-157. doi: 10.1016/j.gie.2019.02.030. Epub 2019 Mar 5. PMID 30849396
- [Background] Karstensen JG, Saftoiu A, Brynskov J, Hendel J, Klausen P, Cartana T, Klausen TW, Riis LB, Vilmann P. Confocal laser endomicroscopy: a novel method for prediction of relapse in Crohn's disease. Endoscopy. 2016 Apr;48(4):364-72. doi: 10.1055/s-0034-1393314. Epub 2015 Nov 19. PMID 26583952
- [Background] Kiesslich R, Duckworth CA, Moussata D, Gloeckner A, Lim LG, Goetz M, Pritchard DM, Galle PR, Neurath MF, Watson AJ. Local barrier dysfunction identified by confocal laser endomicroscopy predicts relapse in inflammatory bowel disease. Gut. 2012 Aug;61(8):1146-53. doi: 10.1136/gutjnl-2011-300695. Epub 2011 Nov 24. PMID 22115910
- [Background] Shavrov A, Kharitonova AY, Davis EM, Claggett B, Morozov DA, Brown DK, Shavrov AA, Liu JJ. A Pilot Study of Confocal Laser Endomicroscopy to Predict Barrier Dysfunction and Relapse in Pediatric Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):873-8. doi: 10.1097/MPG.0000000000001022. PMID 26513619
- [Background] Buchner AM, Wallace MB. Endomicroscopy and Molecular Tools to Evaluate Inflammatory Bowel Disease. Gastrointest Endosc Clin N Am. 2016 Oct;26(4):657-68. doi: 10.1016/j.giec.2016.06.002. Epub 2016 Aug 16. PMID 27633594
- [Background] Abramson O, Durant M, Mow W, Finley A, Kodali P, Wong A, Tavares V, McCroskey E, Liu L, Lewis JD, Allison JE, Flowers N, Hutfless S, Velayos FS, Perry GS, Cannon R, Herrinton LJ. Incidence, prevalence, and time trends of pediatric inflammatory bowel disease in Northern California, 1996 to 2006. J Pediatr. 2010 Aug;157(2):233-239.e1. doi: 10.1016/j.jpeds.2010.02.024. Epub 2010 Apr 18. PMID 20400099
- [Background] Kappelman MD, Moore KR, Allen JK, Cook SF. Recent trends in the prevalence of Crohn's disease and ulcerative colitis in a commercially insured US population. Dig Dis Sci. 2013 Feb;58(2):519-25. doi: 10.1007/s10620-012-2371-5. Epub 2012 Aug 29. PMID 22926499